CLINICAL TRIAL: NCT01709669
Title: The Impact of Gratitude on Biology and Behavior in Persons With Heart Disease
Acronym: GRACE
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director, Blake 11, Massachusetts General Hospital
Other Study IDs: 2012P001191
Record Dates: First submitted 2012-09-21; First posted 2012-10-18 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-03

CONDITIONS: Myocardial Infarction; Unstable Angina
Keywords: acute coronary syndrome; gratitude; health behavior; myocardial infarction; unstable angina
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Acute Coronary Syndrome; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Analyzed Blood Samples:
  Subjects will have a blood draw for the following biological factors that are important to cardiac health and may be modified by psychological states: Inflammation will be measured via interleukin-6 (IL-6) and high sensitivity C-reactive protein (hsCRP), soluble intercellular adhesion molecule-1 (sICAM-1), tumor necrosis factor alpha (TNF-α), and overall cardiac prognosis will be assessed using N-terminal pro-brain natriuretic peptide (NT-proBNP). A total of 15 ml/cc of blood will be drawn (this is equivalent to 3 tablespoons of blood).
  Retained Blood Samples:
  Given that additional, more sensitive/critical markers of cardiac outcomes may be identified in the near future, participants will be given the option to allow us to store their blood samples for additional biomarker analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolling by invitation

SUMMARY:
Overall, the investigators aim to recruit 150 subjects during their hospitalization for an acute coronary syndrome (ACS). At two weeks post-ACS, the investigators will assess levels of gratitude and optimism, draw blood for baseline levels of biomarkers, gather baseline information about health behaviors critical to cardiac health, and obtain baseline measures of symptoms and function. Finally, the investigators will repeat assessments of biomarkers, behavior, and function at 6 months to allow us to assess the impact of gratitude and optimism on these outcomes; the investigators will also have an objective measure of physical activity via accelerometer (step counter) at 6 months.

Specific Aim #1: To prospectively assess the association between gratitude/optimism 2 weeks after ACS and improvement in biological markers of cardiac health at 6 months post-ACS.

Hypothesis: Higher levels of gratitude/optimism at 2 weeks will be associated with greater reductions in levels of biomarkers associated with negative heart health between 2 weeks and 6 months.

Specific Aim #2 (*primary aim*): To assess the association between gratitude/optimism 2 weeks after ACS and subsequent adherence to health behaviors known to improve post-ACS prognosis at 6 months.

Hypothesis: Higher levels of gratitude/optimism at 2 weeks will be associated with greater amounts of physical activity (measured by accelerometer) at 6 months (primary study outcome measure), and greater improvements in self-reported adherence to health behaviors (activity, diet, and medication) between 2 weeks and 6 months.

Specific Aim #3: To assess the association between gratitude/optimism at 2 weeks and non-elective cardiac rehospitalizations (and other clinical outcomes) at 6 months.

Hypothesis: Higher levels of gratitude/optimism at 2 weeks will be associated with greater improvements in depression, health-related quality of life, function, cardiac symptoms, and possibly readmissions, between 2 weeks and 6 months.

DETAILED DESCRIPTION:
Enrollment Patients will be enrolled during their acute admission for an ACS. At this visit, patients will be introduced to the study and given a follow-up study visit at the MGH Heart Center 2 weeks following their ACS. We will also ask them about their physical activity levels in the time before their ACS.

On the date of enrollment, study staff will estimate baseline physical activity using the Stanford 7-day Physical Activity Recall Scale (PAR). Additionally, contact information (address, phone number, email) will be obtained from the subject along with his/her social security number in order to provide a check for compensation.

Initial Evaluation:

After enrollment, subjects will have a visit 2 weeks post-ACS in the MGH Heart Center. Several procedures will occur during this visit.

1. Baseline assessments. Subjects will complete self-report measures to assess the following:

   * Gratitude will be assessed using the Gratitude Questionnaire-6 (GQ-6). The GQ-6 is a brief, validated six-item measure of dispositional gratitude.
   * Optimism will be measured using the Life Orientation Test-Revised (LOT-R), a short 6-item rating scale.
   * Baseline adherence to health behaviors will be measured using items from the MOS Specific Adherence Scale (SAS) that ask about diet and medication adherence.
   * Baseline medical and functional status will be measured using the MOS Short Form-12 (SF-12). The SF-12 is a cardiac symptom scale adapted from the Women and Ischemia Syndrome Evaluation (WISE) study, and the Duke Activity Symptom Index (DASI) for function.
   * Depression will be measured using the Patient Health Questionnaire-9,which is a 9-item scale.
   * Anxiety will be measured using the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS-A). The HADS-A is a 7-item scale.
2. Biomarker collection. Subjects will also have a single blood draw (2 tablespoons or 10 ml/cc) for the following biological factors that are important to cardiac health and may be modified by psychological states. A total of 15 ml/cc of blood will be drawn.
3. Chart review for baseline variables. We will review subjects electronic medical record to gather data on sociodemographic variables (age, gender), medical information (severity of initial ACS), and overall cardiac function.

3 month phone call:

Three months after enrolling in the study, we will call participants to help them test the accelerometer. We will also schedule their 6-month study visit and repeat all self-report measures. Finally, we will remind them to wear the accelerometer for 14 days prior to their 6-month visit and record their physical activity each day for 14 days. We will schedule this call at a convenient time for the participant (on a weekday, weeknight, or weekend).

Provision of accelerometer:

One month before their six-month visit, we will mail the Pebble uniaxial accelerometer (Fitlinxx, Shelton, CT) to the participant, along with an instruction sheet and technical support contact information. We will contact subjects shortly after to make sure the accelerometer arrived, and we will have them wear the devices for several days to ensure that there are no troubles with fit, operation, or remembering to use the devices.

6 month assessment:

Finally, subjects will return to the MGH Heart Center Clinic 6 months post-ACS. At this assessment, we will repeat all self-report measures, collect accelerometers, draw blood (2 tablespoons or 10 ml/cc) for biomarkers, and inquire about readmissions since enrollment. We will gather additional information about readmissions from participants' physicians and medical records for this exploratory outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to cardiac units at MGH with a primary admission diagnosis of ACS (eligible patients must meet World Health Organization criteria for myocardial infarction or criteria for unstable angina [new-onset angina within 2 months, exacerbation of previous angina with rest pain or with minimal exercise, or angina within 2 weeks of MI]). ACS diagnosis will be clarified with the inpatient care team and adjudicated by co-investigator cardiologist Dr. Januzzi as needed.

Exclusion Criteria:

* 'Periprocedural' ACS (ACS that occurs in the setting of another medical procedure; such events may occur in the absence of structural heart disease and likely represent a different pathophysiology, course and prognosis than those with 'endogenous' ACS).
* Conditions likely to alter biomarkers of interest (renal failure requiring hemodialysis, inflammatory disease [e.g., systemic lupus erythematosus])
* Condition likely to lead to death within 6 months (e.g. cancer).
* Inability to complete physical activity due to unrelated medical condition (e.g., severe arthritis)
* Inability to complete self-report evaluations due to inability to speak or write in English or due to cognitive deficits (assessed using an established six-item screen).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Ellison Cardiac Care Units at Massachusetts General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Intake and 6 months after ACS
  Subjects' level of physical activity as measured by an activity recall log and number of steps taken over a two week period measured by an accelerometer.

SECONDARY OUTCOMES:
Biomarkers | 2 weeks and 6 months after ACS
  Levels of inflammation (IL-6, hsCRP, sCAM-1, TNF-α) and overall cardiac prognosis (NT-proBNP)
Readmissions (cardiac and all-cause) | 6 months after ACS
  Non-elective readmissions for cardiac and all causes, ascertained by patient report, report of medical providers, and review of medical records.

OTHER OUTCOMES:
Depression | 2 weeks, 3 months, and 6 months
  Patient Health Questionnaire-9 (PHQ-9)
Anxiety | 2 weeks, 3 months, and 6 months
  Hospital Anxiety and Depression Scale Anxiety Subscale (HADS-A)
Health-Related Quality of Life | 2 weeks, 3 months, and 6 months
  MOS Short Form-12 (SF-12)
Function | 2 weeks, 3 months, and 6 months
  Duke Activity Symptom Index (DASI)
Cardiac Symptoms | 2 weeks, 3 months, and 6 months
  A cardiac symptom scale adapted from the Women and Ischemia Syndrome Evaluation (WISE) study
Adherence to Medical Recommendations | 2 weeks, 3 months, and 6 months
  The MOS Specific Adherence Scale (SAS)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Huffman, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Millstein RA, Celano CM, Beale EE, Beach SR, Suarez L, Belcher AM, Januzzi JL, Huffman JC. The effects of optimism and gratitude on adherence, functioning and mental health following an acute coronary syndrome. Gen Hosp Psychiatry. 2016 Nov-Dec;43:17-22. doi: 10.1016/j.genhosppsych.2016.08.006. Epub 2016 Aug 30. PMID 27796252
- [Derived] Celano CM, Beale EE, Beach SR, Belcher AM, Suarez L, Motiwala SR, Gandhi PU, Gaggin H, Januzzi JL Jr, Healy BC, Huffman JC. Associations Between Psychological Constructs and Cardiac Biomarkers After Acute Coronary Syndrome. Psychosom Med. 2017 Apr;79(3):318-326. doi: 10.1097/PSY.0000000000000404. PMID 27749683
- [Derived] Huffman JC, Beale EE, Celano CM, Beach SR, Belcher AM, Moore SV, Suarez L, Motiwala SR, Gandhi PU, Gaggin HK, Januzzi JL. Effects of Optimism and Gratitude on Physical Activity, Biomarkers, and Readmissions After an Acute Coronary Syndrome: The Gratitude Research in Acute Coronary Events Study. Circ Cardiovasc Qual Outcomes. 2016 Jan;9(1):55-63. doi: 10.1161/CIRCOUTCOMES.115.002184. Epub 2015 Dec 8. PMID 26646818